CLINICAL TRIAL: NCT05455892
Title: Analysis of Mortality, Gravity Predictive Factors and Evolution of Clinical Characteristics of Older Patients Hospitalized for COVID-19 in Short Geriatric Services.
Brief Title: Mortality, Gravity Predictive Factors and Clinical Evolution of Older COVID-19 Patients in Short Geriatric Services.
Acronym: GERICOVID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: AGORA n°36
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: ELDERLY; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elder patients hospitalized for COVID-19 in geriatric short stay units.: All patients over 70 years of age, with a positive Polymerase Chain Reaction or a high presumption of COVID-19, hospitalized in short geriatric units in University Hospital of Lyon, who agree with retrospective collection of their clinical datas.
  Interventions: Other: Clinical data collection during hospitalization in short geriatric units.

INTERVENTIONS:
Other: Clinical data collection during hospitalization in short geriatric units. — Retrospective clinical data collection, at time of infection and 10 days later. Correlation between mortality and gravity. Identification of predictive mortality factors such as frailty, preexisting comorbidities, complications and treatments. Description of medical prescription evolutions.

SUMMARY:
Since the beginning of the year 2020, clinical characteristics of a new disease as the global COVID-19 epidemic has spread in France. People over 70 years of age are the more concerned by this virus in proportion and in gravity with some atypical first symptoms compared to younger patients. Evolution of the disease is variable from forms with few symptoms to severe forms sometimes quickly lethal.

GERICOVID LYON is a descriptive analysis of all patients over 70 years of age hospitalised for COVID-19 in short geriatric unities of University Hospital of Lyon This study will allow more comprehension about COVID-19 in older people. The role of predictive factors, pre-existing comorbidities and the nature and frequency of complications in a short period will be investigate. Treatments practices will be analysed too.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 70 years of age.
* Patient hospitalized in short geriatric units in University Hospital of Lyon.
* Patient diagnosed with COVID-19 (positive Polymerase Chain Reaction or a high presumption of COVID-19 based on clinical and/or scannographic evidence).
* Patient Informed and non-opposed to the research (Patient informed of the study by his medical doctor during hospitalization or by post, thanks to a generic information sheet dedicated to COVID-19 researches).

Exclusion Criteria:

* Patient opposed to the research.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study was proposed to all patients over 70 years of age, with a positive Polymerase Chain Reaction or a high presumption of COVID-19, hospitalized in short geriatric units in University Hospital of Lyon between 1er March 2020 and 30th June 2020.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality rate. | During patient hospitalization, an average of 10 days.
  Observed mortality rate will be presented with its 95% confidence interval.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Service de gériatrie aigue de l'hôpital de la Croix Rousse. Hospices Civils de Lyon, Caluire-et-Cuire, Rhone
  - Service de gériatrie aigue de l'hôpital Edouard Herriot, Pavillon T. Hospices Civils de Lyon, Lyon, Rhone
  - Service de gériatrie aigue de l'hôpital Edouard Herriot. Hospices Civils de Lyon, Lyon, Rhone
  - Service de gériatrie aigue de l'hôpital Lyon Sud. Hospices Civils de Lyon, Pierre-Bénite, Rhone
  - Service de gériatrie aigue de l'hôpital des Charpennes. Hospices Civils de Lyon, Villeurbanne, Rhone

IPD SHARING:
Plan to Share IPD: Undecided